CLINICAL TRIAL: NCT07263633
Title: Additive Versus Subtractive Manufacturing Techniques of Custom-Made Plates for the Fixation of Interforaminal Mandibular Fractures:A Randomized Controlled Trial
Brief Title: Additive Versus Subtractive Manufacturing Techniques of Custom-Made Plates for the Fixation of Interforaminal Mandibular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, FARIS INAD S ALANAZI, Principal Investigator, Master's Student, Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TANTAOMSF-IFMF-149
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Anterior Mandibular Fracture
Keywords: Additive; Subtractive; Custom-Made Plates; Interforaminal; Mandibular; Fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- additive plating group (Experimental): Additive manufacturing typically describes any process where material is gradually added, layer by layer, to form a final product. The term is often used interchangeably with 3D printing and rapid prototyping, although rapid prototyping can also involve other techniques beyond additive methods
  Interventions: Device: additive plating group
- subtractive plating group (Active Comparator): In subtractive manufacturing, objects are created by progressively removing material from a solid block or sheet through processes such as cutting, drilling, boring, or grinding. While these processes can be performed manually, they are more commonly executed using computer numeric control (CNC). CNC machining is the most widely used subtractive manufacturing process today
  Interventions: Device: subtractive plating group

INTERVENTIONS:
Device: additive plating group — Additive manufacturing is the process of creating parts by joining materials based on 3D model data, typically layer by layer, in contrast to subtractive and formative manufacturing methods. While most of the global activity in additive manufacturing currently involves polymer-based systems, there has been increasing interest and activity in fabricating metallic parts
  Arms: additive plating group
Device: subtractive plating group — In CNC machining, cutting tool removes material to achieve the desired geometry. The process involves using CAD to create the model to be machined and CAM to provide instructions to the CNC machine on how to remove the material. There are three major machining processes for material removal based on 3D models: turning, drilling, and milling. Additional subtractive manufacturing techniques, such as laser cutting, waterjet cutting, electrical discharge machining, and plasma cutting, are typically used for 2D machining
  Arms: subtractive plating group

SUMMARY:
This study aims to compare the mechanical properties, including tensile strength, shear strength, and flexural strength, as well as the clinical outcomes of additive and subtractive manufacturing techniques used to fabricate custom-made plates for the fixation of interforaminal mandibular fractures. A total of 16 patients were included and allocated into two groups: one treated using plates fabricated with the additive manufacturing technique and the other with the subtractive manufacturing technique. Mechanical performance was evaluated using standardized biomechanical testing, while clinical outcomes were assessed during scheduled postoperative follow-up visits. The objective of the study is to determine which fixation approach provides superior biomechanical performance and favorable clinical healing outcomes.

DETAILED DESCRIPTION:
This randomized clinical study included 18 patients who were assessed for eligibility. Two patients were excluded-one did not meet the inclusion criteria and another declined participation-leaving a final sample of 16 patients who were randomly allocated into two equal groups (n=8 per group). All included patients were followed throughout the entire study period, and none were lost to follow-up.

Both study groups demonstrated comparable baseline characteristics with no statistically significant differences regarding age, sex distribution, trauma side, cause of injury, type of fracture, and operative time. All surgical procedures were performed using standardized operative protocols, and postoperative evaluations were conducted at fixed intervals.

Clinical outcomes included wound healing status, postoperative edema, infection, and wound dehiscence. Functional performance was evaluated through maximum mouth opening measurements and patient-reported outcomes involving occlusion and self-chewing ability. Radiographic and mechanical assessments were also performed, including tensile strength, shear strength, and flexural bending tests for the fixation systems used in each group.

Across the follow-up period, both groups showed satisfactory wound healing, absence of infection or dehiscence, progressive improvement in mouth opening, and gradual restoration of occlusal stability and chewing function, with no significant intergroup differences in clinical parameters. Mechanical testing demonstrated significant differences between the two fixation systems.

All collected data were statistically analyzed, and outcomes were reported in accordance with CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Isolated or non-isolated mandibular fractures located between the mental foramina (interforaminal fractures).

Exclusion Criteria:

* Patients with relevant systemic diseases that affect bone healing.
* Comminuted fractures in which it is difficult to fix.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Tensile Strength | After fabrication of the plates (baseline biomechanical assessment)
  Tensile strength will be measured using a universal testing machine (Instron) to evaluate the resistance of each plate to tensile forces according to standardized biomechanical testing protocols.
  Unit of Measure:
  Newton (N)
  Measurement Tool:
  Instron Universal Testing Machine.
Shear Strength | Immediately after fixation (within 24 hours)
  Shear strength will be tested using the Instron universal testing machine to determine the resistance of the plate to shear loading.
  Time Frame:
  After fabrication of the plates (baseline biomechanical assessment)
  Unit of Measure:
  Newton (N)
  Measurement Tool:
  Instron Universal Testing Machine.
Outcome Measure | Immediately after fixation (within 24 hours)
  Title: Overall Mechanical Stability Description: Overall biomechanical stability will be evaluated based on combined tensile, shear results.
  Time Frame: Within 24 hours after surgical fixation Unit of Measure: Stability index (unitless)

SECONDARY OUTCOMES:
Mouth Opening Measurement | 1 week, 2 weeks, 1 month, 3 months, and 6 months after surgery
  Maximum inter-incisal distance will be measured using a digital caliper to assess functional recovery and detect any restrictions.
  Unit of Measure:
  Millimeters (mm)
  Measurement Tool:
  Digital caliper
Wound Healing Score | 1 week, 2 weeks, 1 month, 3 months, and 6 months after surgery
  Wound healing will be assessed using the Landry, Turnbull, and Howley Wound Healing Index, which evaluates tissue color, bleeding on palpation, granulation tissue, and overall appearance.
  Unit of Measure:
  Score (0-5 scale)
  Measurement Tool:
  Landry, Turnbull & Howley Index (clinical scale)
Postoperative Edema Measurement | 1 week, 2 weeks, 1 month, 3 months, and 6 months after surgery
  Edema will be measured using standardized linear facial measurements (tragus-pogonion and gonion-pogonion distances) to quantify postoperative swelling.
  Unit of Measure:
  Millimeters (mm)
  Measurement Tool:
  Facial linear measurement with ruler/caliper.
Postoperative Infection Assessment | 1 week, 2 weeks, 1 month, 3 months, and 6 months after surgery
  Infection will be evaluated using the CDC Surgical Site Infection (SSI) criteria, including redness, swelling, warmth, purulent discharge, fever >38°C, and localized tenderness at the surgical site.Unit of Measure:
  Presence or absence (Yes/No)
  Measurement Tool:
  CDC SSI Diagnostic Criteria (clinical assessment)

CONTACTS AND LOCATIONS:
Overall Officials: FARIS I ALANAZI, Principal Investigator — Faculty of Dentistry, Tanta University; Rafic R Bedir, Principal Investigator — Faculty of Dentistry, Tanta University; Ahmed G Abushahba, Principal Investigator — Faculty of Dentistry, Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No